CLINICAL TRIAL: NCT01805804
Title: Randomized, Placebo Controlled Blinded Study to Assess the Efficacy of Valsartan to Prevent Left Ventricle Remodeling in Patients With Dual Chamber Pacemaker
Brief Title: Valsartan to Prevent Left Ventricle Remodeling in Pacemaker Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recall of some valsartan preparations. 88 patients enrolled and completed the observation. All patients are in continuous observation and are well.
Sponsor: Medical University of Silesia (Other)
Collaborators: Polpharma Pharmaceutical Company (Unknown)
Responsible Party: Principal Investigator, Andrzej Tomasik MD PhD FESC, Doctor, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 01/2012; KNW-1-154/P/2/0 (Other Grant/Funding Number: Medical University of Silesia)
Record Dates: First submitted 2013-03-02; First posted 2013-03-06 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: First Time Dual Chamber Pacemaker Implantation
Keywords: dual chamber pacing, left ventricle remodeling, valsartan
MeSH Terms: conditions — Ventricular Remodeling | interventions — Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo pills to match valsartan tablets administered once daily
  Interventions: Drug: placebo/valsartan
- valsartan 80mg daily (Experimental): Valsartan 80mg tablet once daily
  Interventions: Drug: placebo/valsartan
- valsartan 160mg daily (Experimental): Valsartan 160mg tablet once daily
  Interventions: Drug: placebo/valsartan

INTERVENTIONS:
Drug: placebo/valsartan
  Other Names: Valsartan; Other names:; Diovan; Axudan; Vanatex

SUMMARY:
Dual chamber pacing is known to induce left ventricle remodeling and may eventually lead to heart failure. The investigators aim to test hypothesis that valsartan started immediately after dual chamber pacemaker implantation will prevent left ventricle remodeling in twelve months long follow up in comparison with placebo. Echocardiographic assessment of left ventricle remodeling will be correlated with plasma activity of matrix metalloproteinases and their tissue inhibitors, indices of functional capacity such as plasma level of NTproBNP and distance in meters during six minute walking test.

ELIGIBILITY:
Inclusion Criteria:

* informed written consent
* age ≥ 18 years
* first time pacemaker implantation for trifascicular block, atrioventricular second or third degree block
* left ventricle ejection fraction ≥ 40%

Exclusion Criteria:

* significant valvular heart disease
* ischaemic heart disease requiring further revascularization
* symptomatic hypotension
* orthostatic disorders
* pregnancy, breast feeding, child bearing potential
* previous use of angiotensin receptor blocking agents
* known hypersensitivity to valsartan
* significant liver disorders
* significant renal disorders, including renal artery stenosis
* hyperaldosteronism
* chronic use of nonsteroid antiinflammatory drugs
* chronic use of lithium salts
* Patient's reluctance or disability to obey protocol and/or follow the scheduled visits
* any significant disease to reduce the expected life duration < 12 months
* participation in any other trial within the last 30 days before randomization
* any situation that would put more risk on patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
change in echocardiographically assessed left ventricle dimensions and left ventricle function | baseline and 12 months

SECONDARY OUTCOMES:
change in plasma level of matrix metalloproteinase 9 | baseline and 12 months
change in plasma level of NTproBNP | baseline and 12 months
change in atrial arrhythmia burden assessed from pacemaker memory | baseline and 12 months
change in the rate of occurrence of any major adverse cardiovascular event | 2 weeks, 3 months, 6 months, 9 months and 12 months
change in plasma level of tissue necrosis factor alpha | baseline and 12 months
change in plasma level of tissue inhibitor of matrix metalloproteinase 3 | baseline and 12 months
change in distance walked during six minute walking test | baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Nowalany-Kozielska, MD PhD Associate Professor, Study Director — Medical University of Silesia
Locations (1):
- II Dept. of Cardiology in Zabrze Medical University of Silesia, Zabrze, Upper Silesia, Poland

REFERENCES:
- [Background] Suzuki H, Geshi E, Nanjyo S, Nakano H, Yamazaki J, Sato N, Tanaka K, Takano T, Yagi H, Shibata T, Mochizuki S, Katagiri T. Inhibitory effect of valsartan against progression of left ventricular dysfunction after myocardial infarction: T-VENTURE study. Circ J. 2009 May;73(5):918-24. doi: 10.1253/circj.cj-08-0959. Epub 2009 Apr 2. PMID 19346662
- [Background] Miyazaki S, Kasai T, Miyauchi K, Miyazaki T, Akimoto Y, Takagi A, Aihara K, Kawamura M, Suwa S, Kojima S, Sumiyoshi M, Daida H. Changes of matrix metalloproteinase-9 level is associated with left ventricular remodeling following acute myocardial infarction among patients treated with trandolapril, valsartan or both. Circ J. 2010 Jun;74(6):1158-64. doi: 10.1253/circj.cj-09-0412. Epub 2010 Apr 6. PMID 20378999
- [Background] Garcia RA, Brown KL, Pavelec RS, Go KV, Covell JW, Villarreal FJ. Abnormal cardiac wall motion and early matrix metalloproteinase activity. Am J Physiol Heart Circ Physiol. 2005 Mar;288(3):H1080-7. doi: 10.1152/ajpheart.00860.2004. Epub 2004 Oct 14. PMID 15486029
- [Derived] Tomasik A, Jachec W, Wojciechowska C, Kawecki D, Bialkowska B, Romuk E, Gabrysiak A, Birkner E, Kalarus Z, Nowalany-Kozielska E. Randomized placebo controlled blinded study to assess valsartan efficacy in preventing left ventricle remodeling in patients with dual chamber pacemaker--Rationale and design of the trial. Contemp Clin Trials. 2015 May;42:239-43. doi: 10.1016/j.cct.2015.03.015. Epub 2015 Apr 7. PMID 25858003